CLINICAL TRIAL: NCT04658290
Title: Prevalence of Obstructive Sleep Apnea (OSA) and the Association With Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: SleepBrain_2019
Record Dates: First submitted 2020-08-31; First posted 2020-12-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea; Cognitive Impairment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed to carry out an epidemiology study investigating the prevalence of obstructive sleep apnea (OSA) and the association with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Have stability of at least 4 weeks on permitted medications (i.e. medications known not to affect sleep architecture or circadian rhythms).

Exclusion Criteria:

* Suspected dementia or a score of <24 on the mini-mental state examination
* A diagnosis of neurological disorders (e.g. Parkinson's Disease, Epilepsy, Multiple Sclerosis)
* Psychiatric disorders including current major depression; bipolar disorder; schizophrenia
* Other known clinically significant sleep disorders (e.g. narcolepsy)
* Been currently receiving CPAP or bi-level pressure for OSA

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects are recruited from the Brain Health Longitudinal Study which was launched in July 2019. Up to 5000 subjects aged 40-74 years without a confirmed brain disorder. Participants will be assigned to undergo a portable at-home sleep study which records the airflow, heart rate, body position and oxygen saturation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-29 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of subjects having apnea-hypopnea index of more than 5 | 1 year

SECONDARY OUTCOMES:
incidence of cerebrovascular disease | 5 years
Montreal Cognitive Assessment | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong, Hong Kong, Please Select, Hong Kong